# Statistical Analysis Plan

Protocol Number: MCI-186-J25

A Randomized, Single-Blind, Placebo-Controlled,
Three-Way Crossover Study to Evaluate the Effect of
MCI-186 at Therapeutic and Supra-Therapeutic
Doses on the QT/QTc Interval in Healthy Subjects

Version Number: 2.0 Date: January 25, 2019

NCT number: NCT04029090

## STATISTICAL ANALYSIS PLAN

Protocol No.

MCI-186-J25

Protocol Title

A Randomized, Single-Blind, Placebo-Controlled, Three-Way Crossover Study to Evaluate the Effect of MCI-186 at Therapeutic and Supra-Therapeutic Doses on the QT/QTc Interval in Healthy Subjects

Version History

Version 1.0 First approved version / 16 January, 2019

Version 2.0 Final approved version / 25 January, 2019

Author

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation. Protocol No. MCI-186-J25 Date: 25 January, 2019

## APPROVAL FORM

The approval signatories below have reviewed this Statistical Analysis Plan (SAP) and agreed on the planned analyses defined in this document.

| MTPC Statistics Approve | | [MTPC-STATH] |
|-------------------------|----------|----------------|
| | Date: | Signature: |
| | -<br>- | . <del>.</del> |
| MTR@ Pharmacokinetics | Approver | [MTPC-STATH] |
| | Date: | Signature: |
| | _ | |
| | | · |

## TABLE OF CONTENTS

| 1. | INT | RODUCTION | 9 |
|----|-----|--------------------------------------------------|---|
| | 1.1 | Study Design | 9 |
| | 1.2 | Schedule of Study Procedures | 9 |
| 2. | STU | DY OBJECTIVES AND ENDPOINTS1 | 1 |
| | 2.1 | Study Objectives | 1 |
| | | 2.1.1 Primary objective | 1 |
| | | 2.1.2 Secondary objectives | 1 |
| | | 2.1.3 Primary endpoint | 1 |
| | | 2.1.4 Secondary endpoints | 1 |
| | | 2.1.5 Exploratory endpoints | 1 |
| 3. | PLA | NNED ANALYSES1 | 1 |
| 4. | ANA | LYSIS POPULATION(S)1 | 2 |
| 5. | GEN | ERAL CONSIDERATIONS1 | 2 |
| | 5.1 | Subjects Composition | 2 |
| | 5.2 | Analysis Time Window for Visits | 2 |
| | 5.3 | Handling of data for pharmacokinetic assessments | 4 |
| | 5.4 | Number of Digits to Report | 4 |
| | 5.5 | Significance level and confidence level1 | 4 |
| | 5.6 | Descriptive statistics values to calculate | 4 |
| | 5.7 | Derived variables | 4 |
| 6. | SAN | IPLE SIZE AND POWER CONSIDERATIONS1 | 5 |
| 7. | STA | TISTICAL METHODOLOGY1 | 6 |
| | 7.1 | Disposition of Subjects | 6 |
| | 7.2 | Demographic and Other Baseline Characteristics | 6 |
| | 7.3 | Medical History | 6 |
| | 7.4 | Prior and Concomitant Medications1 | 6 |

8.

9.

| 7.5 | Study | Drug Exposure | 17 |
|-----|----------|-----------------------------------------------------|----|
| 7.6 | Treatm | nent Compliance | 17 |
| 7.7 | Statisti | ical/Analytical issues | 17 |
| | 7.7.1 | Adjustments of covariates | 17 |
| | 7.7.2 | Handling of Dropouts or Missing Data | 17 |
| | 7.7.3 | Interim Analyses and Data Monitoring | 17 |
| | 7.7.4 | Multicentre Studies | 17 |
| | 7.7.5 | Multiple Comparison/Multiplicity | 17 |
| | 7.7.6 | Use of an "Efficacy Subset" of Patients | 17 |
| | 7.7.7 | Active-Control Studies Intended to Show Equivalence | 18 |
| | 7.7.8 | Examination of Subgroups | 18 |
| | 7.7.9 | Handling of Routine safety laboratory tests Values | 18 |
| | 7.7.10 | Handling of re-examination data | 18 |
| 7.8 | Pharm | acokinetic Assessments | 18 |
| | 7.8.1 | Analysis of Individual Plasma Concentrations | 18 |
| | 7.8.2 | Analysis of Pharmacokinetic Parameters | 19 |
| 7.9 | Safety | Assessments | 19 |
| | 7.9.1 | Adverse Events | 19 |
| | 7.9.2 | Routine safety laboratory tests | 20 |
| | 7.9.3 | Vital Signs and Body Weight | 21 |
| | 7.9.4 | Routine safety 12-lead ECG | 21 |
| | 7.9.5 | Physical Examinations | 21 |
| | 7.9.6 | Withdrawals | 22 |
| | 7.9.7 | Other Safety Assessments | 22 |
| CH | ANGES | FROM THE PROTOCOL | 22 |
| DA | TA NO | Γ SUMMARISED OR PRESENTED | 22 |
| DEI | ED ENI | TEQ. | 22 |

| Statistical Analysis Plan |
|---------------------------------------|
| Mitsubishi Tanabe Pharma Corporation. |

| 11. VALIDATIONS | 22 |
|---|---|
| 12. LISTINGS, TABLES AND FIGURES | 23 |
| 12.1 Listings | 23 |
| 12.2 Tables | 23 |
| 12.3 Figures | 24 |
| 13. REVISION HISTORY FOR SAP AMENDMENTS | 25 |
| APPENDIX 1 – CALCULATION OF PHARMACOKINETIC PARAMETER USING NON-COMPARTMENTAL ANALYSIS | 26 |
| APPENDIX 2 – CALCULATION OF PHARMACOKINETIC PARAMETER USING COMPARTMENTAL ANALYSIS | 29 |

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation. Protocol No. MCI-186-J25 Date: 25 January, 2019

## Abbreviations

WHO-DD:

| AE | : | adverse event |
|-------|----|----------------------------------------------|
| BLQ | : | below limit of quantification |
| BMI | : | body mass index |
| CV | : | coefficient of variation |
| DBL | : | database lock |
| DP | : | decimal places |
| ECG | : | electrocardiogram |
| IAO | : | International agreed order |
| IMP | :. | investigational medicinal product |
| LLOQ | : | lower limit of quantification |
| MedDR | A: | Medical Dictionary for Regulatory Activities |
| PK | : | pharmacokinetics |
| PT | : | preferred term |
| QC | : | quality control |
| SAP | : | statistical analysis plan |
| SAE | : | serious adverse event |
| SD | : | standard deviation |
| SOC | : | system organ class |
| TEAE | : | treatment emergent adverse event |

World Health Organization Drug Dictionary

| Parameters | Unit | Definitions |
|---|---|---|
| α | 1/h | Elimination rate constant of the α-phase |
| AUC <sub>0-last</sub> | h*ng/mL | Area under the concentration-time curve from time zero to the last quantifiable concentration time point |
| AUC <sub>0-24h</sub> | h*ng/mL | Area under the concentration-time curve from time zero to 24 |
| AUC <sub>0-∞</sub> | h*ng/mL | Area under the concentration-time curve from time zero to infinity |
| AUC% <sub>ex</sub> | % | Area under the plasma concentration-time curve extrapolated from the last quantifiable concentration time point to infinity in % of the total $AUC_{0-\infty}$ |
| β | 1/h | Elimination rate constant of the β-phase |
| CL | L/h | Total clearance |
| C <sub>max</sub> | ng/mL | Maximum plasma concentration |
| γ | 1/h | Elimination rate constant of the γ-phase |
| k <sub>21</sub> | 1/h | Transfer rate constant from peripheral (2) to central (1) compartment |
| k <sub>31</sub> | 1/h | Transfer rate constant from peripheral (3) to central (1) compartment |
| k <sub>el</sub> | 1/h | Elimination rate constant from the central compartment in compartmental analysis |
| Lower limited of $\lambda_z$ | h | Lower data point used for the estimation of $\lambda_z$ |
| MRT | h | Mean residence time |
| Number of $\lambda_z$ points | - | Number of data point used for the estimation of $\lambda_z$ |
| A | ng/mL | Zero-time intercept for α-phase |
| В | ng/mL | Zero-time intercept for β-phase |
| С | ng/mL | Zero-time intercept for γ-phase |
| $\lambda_{z}$ | 1/h | Elimination rate constant in non-compartmental analysis |
| t <sub>1/2</sub> | h | Terminal elimination half-life in plasma concentration-time course |
| t <sub>1/2α</sub> | h | Half-life at α-phase |
| t <sub>1/2β</sub> | h | Half-life at β-phase |
| t <sub>1/2γ</sub> | h | Half-life at γ-phase |
| t <sub>max</sub> | h | Time of maximum plasma concentration after administration |

| | | List of PK Parameters |
|---|---|---|
| Upper limited of $\lambda_z$ | h | Upper data point used for the estimation of $\lambda_z$ |
| $V_1$ | L | Volume of the central compartment |
| V <sub>SS</sub> | L | Volume of distribution at Steady State |
| V <sub>z</sub> | L | Volume of distribution during terminal phase |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) is based on the final protocol dated 29 August 2018. The plan covers statistical analysis plan, tabulations and listings of to evaluate the effect of MCI-186 at therapeutic and supra-therapeutic doses on the QT/QTc interval in healthy subjects. Holter ECG analysis with the related section of 2 will be performed based on a separate ECG SAP.

The SAP is prepared by The statistical analyses and production of the outputs described in the SAP will be conducted and QC checked by Data Science Department, using SAS® Version 9.2 or higher. The final analyses and outputs will be approved by Mitsubishi Tanabe Pharma Corporation Data Science Department.

### 1.1 Study Design

This is a Phase I, randomized, single-blind, placebo-controlled, three-way crossover single-center study.

Up to 27 healthy male volunteers, aged 20 to 55 years who meet the study criteria will be allocated to 3 treatment sequences of 9 subjects each. In each sequence, subjects will receive a single I.V. dose of MCI-186 as therapeutic or supra-therapeutic dose, or a matching dose of placebo in a fasted state.

The study consists of the following 3 treatments and 3 sequences;

- Treatment A (therapeutic dose of MCI-186): A single dose of 60 mg MCI-186 over 60 min will be intravenously administered.
- Treatment B (supra-therapeutic dose of MCI-186): A single dose of 300 mg MCI-186 over 60 min will be intravenously administered.
- Treatment C (Placebo): A single dose of 0.9% w/v saline over 60 min will be intravenously administered.

| Sequence | Period 1 | Period 2 | Period 3 |
|----------|----------|----------|----------|
| 1 | A | С | В |
| 2 | В | A | C |
| 3 | C | В | Α |

## 1.2 Schedule of Study Procedures

Study assessments are summarized in the time and events schedule in Table 1

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation. Protocol No. MCI-186-J25 Date: 25 January, 2019

Table 1 Time and events schedule

| | | Confinement | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | Screen-<br>ing | | | | | | | | | | Follow-up | | | | | | |
| Study Day | -28 to -3 | -1 | 1 | | | | | | | - | | | | | | 2 | 5-9 |
| Time point in Relation to Start | | | Pre- | | 0.5 | | 75 | 90 | 105 | ٠. | ١., | | | | | | (only |
| of Infusion | | | dose | 0 | h | 1 h | min | min | min | 2 h | 3 h | 4h | 6h | 8h | 12h | 24h | Period 3) |
| Informed consent | X | | ļl | | | | | | | | | | | · | | | |
| Confinement <sup>a</sup> | | <b>&lt;</b> | | | <del> </del> | | | | | | | | | | | > | |
| Outpatient | X | | l | | | <u> </u> | | | | | | | | | | | X |
| Demography & medical history | X | <u> </u> | ļ! | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | X | | ļ | I | | | | | | | | | <u></u> | | |
| Randomization | | | X | | | | | | | | | | <u> </u> | | | | |
| Physical examination | X | X <sup>b</sup> | X <sup>b</sup> | | | Χ <sup>b</sup> | | | | | | | | | | X <sup>b</sup> | X |
| Weight | X | X | | | ļ | | | | | | | | | | | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| BMI | X | X | | | | | | | | | | | | | | | |
| Vital signs <sup>c</sup> | X | X | X | | | X | | | | | l | | | | | X | X |
| Routine safety 12-lead ECGd | Χ° | X | X | | | X | | | | | | | | | | X | X |
| Continuous 12-lead Holter (PD ECGs extracted in triplicate) <sup>f</sup> | | | Xº | | X | х | х | x | х | х | х | х | х | X | х | х | |
| Drugs of abuse & alcohol test | X | X | | | | | | | | | | | | L | | | |
| Hematology, biochemistry, coagulation & urinalysis | X | х | | | | | | | | | | | | | | х | х |
| Serology | X | | | | | | | | | | <u> </u> | | | | | | |
| IMP administration (infusion) | | | | < | | > | | | | | | | | | | | |
| PK sampling (blood)h | | | X | | X | X | X | X | X | X | X | X | X | X | X | X | |
| Adverse events | <b>&lt;</b> | <del> </del> | + | | | <del> </del> | | <del> </del> | | | | | <u> </u> | | | | > |
| Concomitant medications | <b>&lt;</b> | ļ | + | | | ļ | | ∔ <b>-</b> ∙ | <del> </del> | <b></b> | <del> </del> | | <b>+</b> - | <del> </del> | <u> </u> | | <del>&gt;</del> |

Concomitant medications

a: Subjects will be admitted 3 times to the study center (on Day -1 in each period) and discharged in the morning of Day 2 in each period. b: Abbreviated physical exam

b: Abbreviated physical exam

c: Blood pressure, pulse rate and body temperature

d: Using conventional bedside equipment

e: Routine safety ECG in triplicate at Screening only

f: Mandatory rest from 10 minutes prior to until 5 minutes after each timepoint

g: Predose at -45, -30 and -15 minutes

h: No sooner than 5 minutes after associated PD ECG timepoint

#### 2. STUDY OBJECTIVES AND ENDPOINTS

In this SAP, the analyses with underline are not planed.

## 2.1 Study Objectives

#### 2.1.1 Primary objective

• To evaluate the effect of MCI-186 on the QT interval corrected for heart rate using Fridericia's formula (QTcF)

## 2.1.2 Secondary objectives

- To evaluate the PK profile of MCI-186
- To evaluate the effect of MCI-186 on other 12-lead ECG intervals
- To evaluate the safety and tolerability of MCI-186

## 2.1.3 Primary endpoint

• Relationship of change from baseline in QTcF (ΔQTcF) with placebo adjustment (ΔΔQTcF) and concentration of MCI-186

#### 2.1.4 Secondary endpoints

- Assessment of HR, PR interval, QRS interval, and QTcF by timepoint
- Categorical outliers for QTcF interval (absolute value and change from baseline) and other 12-lead ECG parameters
- Incidence of abnormalities in ECG morphology
- PK parameters of MCI-186
- Incidence of adverse events (AEs) and serious adverse events (SAEs), vital signs, safety 12-lead ECG variables, laboratory tests and physical examination

## 2.1.5 Exploratory endpoints

Not applicable in the study.

#### 3. PLANNED ANALYSES

This study was planned to evaluate the effect of MCI-186 at therapeutic and supra-therapeutic doses on the QT/QTc interval in healthy subjects.

The statistical analyses will be performed after database lock(DBL). Interim analysis will not be carried out.

# 4. ANALYSIS POPULATION(S)

The statistical analysis will be based on the following defined populations:

• Safety population includes all randomized subjects who received at least one dose of IMP.

Protocol No. MCI-186-J25 Date: 25 January, 2019

• PK population includes all randomized subjects who received at least one dose of IMP and who have at least one post-dose value of plasma concentration without important Protocol deviations which may affect the PK of the IMP.

For cases that subjects were not adopted in the PK analysis set, all PK data will be rejected and no parameters will be calculated. Furthermore, for cases that subjects adopted in the PK analysis set and partial data not being adopted, PK parameters will be calculated from only the adopted data.

The acceptance or rejection of each analysis population will be treated based on the results of the data review meeting on as follows.

Safety analysis set: No subject is excluded from analysis.

PK analysis set: No subject is excluded from analysis.

#### 5. GENERAL CONSIDERATIONS

#### 5.1 Subjects Composition

- Treatment A (therapeutic dose of MCI-186):
   A single dose of 60 mg MCI-186 over 60 min will be intravenously administered.
- Treatment B (supra-therapeutic dose of MCI-186):
  A single dose of 300 mg MCI-186 over 60 min will be intravenously administered.
- Treatment C (Placebo):
   A single dose of 0.9% w/v saline over 60 min will be intravenously administered.

#### 5.2 Analysis Time Window for Visits

1) Analysis time windows for blood sampling for PK measurements are as follows.

| Pre-dose | Before dosing |
|---|---|
| 0.5 h after dosing | Scheduled time + 5 to 7 minutes |
| 1 h after dosing | Following completion of dosing + 5 to 7 minutes |
| 75 min, 90 min and 105 min after dosing | Scheduled time + 5 to 7 minutes |
| 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 24 h after dosing | Scheduled time + 5 to 10 minutes |

## 2) Analysis time windows for vital signs and safety 12-lead ECG are as follows.

| Screening (Day -28 to Day -3) | Not specified |
|---|---|
| Hospitalization (Day -1) | Not specified |
| Before dosing (Day 1) | From the time of waking up until the time when Holter ECG rest was secured (45 minutes before starting administration) |
| 1 h after dosing (Day 1) | Scheduled time ± 20 minutes |
| 24 h after dosing (Day 2) | From wake-up to scheduled time + 1 hour (25 hours after start of administration) |
| Follow-up (Day $7 \pm 2$ days)* | Not specified |

<sup>\*:</sup> Period 3 only

## 3) Analysis time windows for physical examinations are as follows.

| Screening (Day -28 to Day -3) | Not specified |
|---|---|
| Hospitalization (Day -1) | Not specified |
| Before dosing (Day 1) | From the time of waking up until the time when Holter ECG rest was secured (45 minutes before starting administration) |
| 1 h after dosing (Day 1) | Scheduled time + 1 hour 30 minutes |
| 24 h after dosing (Day 2) | From wake-up to scheduled time + 1 hour (25 hours after start of administration) |
| Follow-up (Day 7 ± 2 days)* | Not specified |

<sup>\*:</sup> Period 3 only

# 4) Analysis time windows for blood and urine sampling at the safety laboratory tests are as follows.

| Screening (Day -28 to Day -3) | Not specified |
|---|---|
| Hospitalization (Day -1) | Not specified |
| 24 h after dosing (Day 2) | Blood sampling: From getting up to before breakfast Urine collection: From getting up to before breakfast |
| Follow-up (Day 7 ± 2 days)* | Not specified |

<sup>\*:</sup> Period 3 only

## 5.3 Handling of data for pharmacokinetic assessments

The allowable ranges for the collection of blood samples for the measurement of the plasma drug concentrations are shown in Section 5.2. Only valid PK data will be included in the summary tables or figures. PK data that are considered "invalid" or "abnormal" will be flagged in the listing. The PK data handling will be confirmed during data review.

## 5.4 Number of Digits to Report

Statistical analysis variables, statistics to be calculated and number of digits to report are as follows.

| Routine safety laboratory tests Physical examinations Routine safety 12-Lead ECG | Mean, SD, median | Report to one extra digit plus the determined/specified digits |
|---|---|---|
| Demography, body weight, height, BMI | Minimum, maximum | Report to the determined/specified digits |
| Pharmacokinetics | Mean, SD, minimum, median, maximum, geometric mean | Report to the determined/specified digits |
| General information | Number of subjects, number of valid observations, number of events, number of cases | Integer |
| | CV%, geometric CV%,<br>Percentages (%) | To the first decimal place |

#### 5.5 Significance level and confidence level

No statistical testing and estimation will be performed.

### 5.6 Descriptive statistics values to calculate

Where appropriate, continuous variables will be summarized descriptively, using the number of observations, mean, SD, median, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages.

#### 5.7 Derived variables

### (1) Definition(s) of baseline(s)

The baseline of vital signs and Routine safety 12-lead ECG is the last valid assessment obtained on or before Day 1 prior to the administration of single-blind IMP by each treatment group (60 mg group, 300 mg group and placebo group).

The baseline of body weight, BMI, and clinical laboratory values will be the value obtained on Day -1.

## (2) Age at informed consent

Age (years) = Year of informed consent - Year of birth

Subtract 1 from the age (years) calculated above, if [Month of informed consent < Month of birth] or [Month of informed consent = Month of birth AND Day of informed consent < Day of birth].

## (3) BMI

 $BMI = Weight [kg] / (Height [m])^2$ 

Height will be the value obtained at screening.

#### (4) Adverse events

The MedDRA version 21.0 will be used as a unified dictionary in the assessment of AEs.

#### (5) Adverse reactions

Adverse reactions are defined as AEs that are determined to have a "Reasonable Possibility" of causal relationship to the IMP.

#### (6) Prior and Concomitant Medications

All medication data will be coded according to the latest version of WHO-DD and Anatomical Therapeutic Chemistry (ATC) classification.

## 6. SAMPLE SIZE AND POWER CONSIDERATIONS

The sample size of 27 subjects of IMP per treatments is not based on a formal power calculation. However, referring to the recent publication<sup>[1]</sup>, even if assuming that is at most 5 msec  $\Delta\Delta QTcF$  in  $C_{max}$  of MCI-186 300 mg as supra-therapeutic dose, 24 subjects of each doses MCI-186 or placebo are considered to be adequate to meet the objectives of the study at power = 80% or higher. In addition, 24 subjects will provide at least 90% power of the upper bound in 90% confidence interval is less than 10 msec, assuming 0 msec  $\Delta\Delta QTcF$  at  $C_{max}$  of MCI-186 60 mg and 300 mg based on simulation using previous studies including MCI-186-E02. Assuming a few drop-out, a total of 27 subjects are planned to be randomized in this study.

## 7. STATISTICAL METHODOLOGY

#### 7.1 Disposition of Subjects

Disposition of subjects will be listed.

- Number and percent of subjects completed and discontinued protocol with its reason will be presented by each sequence (1: A-C-B, 2: B-A-C and 3: C-B-A).
- > Subjects withdrawn will be summarized by reasons for discontinuation.

## 7.2 Demographic and Other Baseline Characteristics

Major demographic and other baseline characteristics will be listed.

For each analysis set, major demographic and other baseline characteristics will be summarized by each sequence (1: A-C-B, 2: B-A-C and 3: C-B-A) and overall. For categorical values, frequency and percentage will be reported. For continuous values, descriptive statistics values (number of subjects, mean, SD, minimum, median, and maximum) will be calculated.

Table. Variables related to demographic and other baseline characteristics

| Category | Variable Data format | |
|---|---|---|
| Subject | Sex (male, female): display without female | Binary |
| background | Age at consent acquisition (years) | Continuous |
| | Race | Categorical |
| | Japanese, Non-Japanese | Binary |
| | Height (cm) | Continuous |
| | Body weight (kg) on Day -1 | Continuous |
| | BMI on Day -1 | Continuous |
| Medical history | | Binary |

#### 7.3 Medical History

All medical history data will be listed.

#### 7.4 Prior and Concomitant Medications

All medication data will be listed.

Prior medication is any medication taken only in the two weeks prior to administration of IMP. Concomitant medication is defined as any medication, other than the IMP, which is taken from the start of IMP infusion to the Follow-up assessment, including prescription, herbal and overthe-counter medications.

Prior and Concomitant medications will be summarized by each treatment group (60 mg group, 300 mg group and placebo group). Incidence tables will be summarized with ATC Level 2 code, text and Drug Code, Drug Name.

The period of Concomitant medications use in each group is as follows.

Period 1: After administration in 1st Treatment to before administration in 2nd Treatment.

Period 2: After administration in 2nd Treatment to before administration in 3rd Treatment.

Period 3: After administration in 3rd Treatment to end of follow up.

## 7.5 Study Drug Exposure

All exposure data will be listed.

## 7.6 Treatment Compliance

All compliance data will be listed.

## 7.7 Statistical/Analytical issues

## 7.7.1 Adjustments of covariates

No statistical testing and estimation will be performed.

## 7.7.2 Handling of Dropouts or Missing Data

Missing data, such as rejected values, will not be imputed.

## 7.7.3 Interim Analyses and Data Monitoring

Not applicable in the study.

## 7.7.4 Multicentre Studies

Not applicable in the study.

## 7.7.5 Multiple Comparison/Multiplicity

No statistical testing and estimation will be performed.

## 7.7.6 Use of an "Efficacy Subset" of Patients

Not applicable in the study.

## 7.7.7 Active-Control Studies Intended to Show Equivalence

Not applicable in the study.

## 7.7.8 Examination of Subgroups

Not applicable in the study.

## 7.7.9 Handling of Routine safety laboratory tests Values

In the case of clinical laboratory test values including equality and inequality sign, exclude equality and inequality sign and use for summarized.

## 7.7.10 Handling of re-examination data

For the re-examination at screening, the examination value of the re-examination at the point closest to date of IMP is adopted.

If there is unscheduled data after the date of IMP, it will be excluded from calculation of summary statistics and frequency aggregation.

#### 7.8 Pharmacokinetic Assessments

### 7.8.1 Analysis of Individual Plasma Concentrations

All measured plasma concentrations will be listed.

Plasma concentrations will be summarized at each scheduled sampling time point by each MCI-186 group (60 mg group and 300 mg group). The following descriptive statistics will be calculated: N (number of subjects), n (number of valid observations), arithmetic mean, SD, CV%, minimum, median, maximum, geometric mean and geometric CV%. Nominal sampling times will be displayed in the summary. For the calculation of the descriptive statistics other than geometric mean and geometric CV%, concentration values reported as BLQ will be set to 0. For the calculation of the geometric mean and geometric CV%, concentration values reported as BLQ will be set to ½ of LLOQ.

CV% and Geometric CV% will be calculated as follows:

$$CV\% = \frac{SD}{arithmetic\ mean} \times 100$$

Geometric CV% = 
$$\left[\exp(\sigma^2) - 1\right]^{1/2} \times 100$$

where  $\sigma$  represents the SD computed on the natural logarithmic transformed concentrations.

To visualize the concentration-time profiles of each MCI-186 group, the following plots will be produced in linear and semi-logarithmic scales:

Statistical Analysis Plan Mitsubishi Tanabe Pharma Corporation.

- 1. Individual subject observed and predicted concentration-time plot with each MCI-186 group (60 mg group and 300 mg group) overlaid in one graph by subject.
- 2. Individual subject observed concentration-time plot overlaid in one graph by each MCI-186 group (60 mg group and 300 mg group).
- 3. Mean observed and predicted concentration-time plot with each MCI-186 group (60 mg group and 300 mg group) overlaid in one graph.
- 4. Mean observed concentration-time plot with each MCI-186 group (60 mg group and 300 mg group) overlaid in one graph.

In the summary tables, arithmetic mean, SD, minimum, median, maximum and geometric mean will be presented with the number of significant digits which individual concentrations are reported. In addition, CV%, and geometric CV% will be presented with 1 decimal place.

## 7.8.2 Analysis of Pharmacokinetic Parameters

All PK parameters will be listed.

The PK parameters will be summarized by each MCI-186 group (60 mg group and 300 mg group). The following descriptive statistics will be calculated: N (number of subjects), n (number of valid observations), arithmetic mean, SD, CV%, minimum, median, maximum, geometric mean and geometric CV%.

For the descriptive statistics, the minimum and maximum will be presented according to following requirement:

- C<sub>max</sub>, A, B, C will be presented with the number of significant digits they are reported with.
- Other PK parameters: will be presented with a fixed number of decimal places for each parameter. The number of decimal places is 2 decimal places corresponding to having 3 significant digits at the minimum by analyte.

Mean, SD, median and geometric mean will be presented with the number of decimals as follows.

- C<sub>max</sub>, A, B, C: will be presented with 4 significant digits.
- Other PK parameters: will be presented with 2 decimal places.

CV% and geometric CV% will be presented with 1 decimal place.

#### 7.9 Safety Assessments

No imputation will be made in case of missing values.

## 7.9.1 Adverse Events

Adverse events will be coded using MedDRA. All AEs for each subject, including multiple occurrences of the same event, will be presented in full in a comprehensive listing including start/stop times, verbatim term, Preferred Term, System Organ Class (SOC), dose level, severity, seriousness, relationship to treatment and outcome will be provided.

Duration of the AE and time to the AE occurrence from start of the IMP will be calculated and presented in days and time.

AE Occurrence from Start of IMP = Date of Onset - Date of Administration +1.

Duration of AE = Date of Resolution - Date of Onset +1.

AEs which start on or after dosing that are expressed or exacerbated are defined as treatment emergent adverse events (TEAEs).

In the tabulations, numbers of subjects with TEAEs will be counted by each treatment group (60 mg group, 300 mg group and placebo group).

The period of AE occurrence in each group is as follows.

- Period 1: After administration in 1st Treatment to before administration in 2nd Treatment.
- Period 2: After administration in 2nd Treatment to before administration in 3rd Treatment.
- Period 3: After administration in 3rd Treatment to end of follow up.

Following summaries of TEAEs will be presented:

- > Summary of TEAEs by SOC and PT
- > Summary of TEAEs by SOC, PT and severity of event
- > Summary of TEAEs by SOC, PT and maximum IMP relationship

Proportion of subjects with any TEAE, subjects with any adverse drug reactions, subjects with any TESAE (Treatment Emergent SAE), subjects with any serious adverse drug reactions, and subjects with any TEAE leading to discontinuation of the study will be summarized.

The summary will be sorted by International Agreed Order (IAO) for SOC and alphabetical order for PT (or by frequency from the highest to the lowest).

For summaries of AEs multiple occurrences of the same event within a subject will be counted once in the summaries by SOC and PT; multiple occurrences of the same event within a subject will be counted once in the maximum intensity category (severe > moderate > mild) and/or maximum drug relationship category (reasonable possibility>no reasonable possibility). If intensity or relationship is found to be missing the most severe occurrence will be imputed for that particular summary.

## 7.9.2 Routine safety laboratory tests

All routine safety laboratory tests parameter will be listed.

Clinical significance of routine safety laboratory tests findings will be evaluated by the Investigator with respect to pre-defined clinically relevant ranges taking into account the Investigator site's normal ranges. The routine safety laboratory tests data will be listed in full with clinically relevant values flagged (L=Lower than normal range, H=Higher than normal range or A=Abnormal if no reference range). A listing of routine safety laboratory tests values will be provided for subjects with any clinical significant findings (list relevant routine safety laboratory tests parameters only).

Lab parameter values and changes from baseline will be summarized descriptively by each treatment group (60 mg group, 300 mg group and placebo group) and analysis visit window. Overall evaluation (Clinical Assessment) for each routine safety laboratory tests will be summarized using frequency and percentage.

Shift tables will present the changes in clinically relevant categories from baseline to each scheduled post-baseline visit. The categories will be qualitative values for Urinalysis (glucose, protein, occult blood, ketone bodies, urobilinogen, erythrocytes, leukocytes, squamous epithelial cells).

#### 7.9.3 Vital Signs and Body Weight

All vital sign and body weight data will be listed.

Vital signs (systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) /body weight values and changes from baseline will be summarized descriptively by analysis visit window. Overall evaluation for vital sign will be summarized using frequency and percentage.

#### 7.9.4 Routine safety 12-lead ECG

All Routine safety 12-lead ECG (heart rate, RR, PR, QRS, QT, QTcF, overall evaluation) parameters and findings will be listed.

Routine safety 12-lead ECG parameter values and changes from baseline will be summarized descriptively by analysis visit window. Overall evaluation for routine safety 12-lead ECG will be summarized using frequency and percentage.

For ECGs, number and percentage of subjects meeting the criteria listed below will be presented:

- > OTcF > 500 msec at time point
- > 500msec >= QTcF > 480 msec at time point
- > 480msec >= QTcF > 450 msec at time point
- > QTcF <= 450 msec at time point
- ➤ Change from baseline in QTcF > 30 msec
- ➤ Change from baseline in QTcF > 60 msec

#### 7.9.5 Physical Examinations

All physical examinations data will be listed.

#### 7.9.6 Withdrawals

All subjects who are withdrawn from the study will be listed.

## 7.9.7 Other Safety Assessments

Not applicable in the study.

## 8. CHANGES FROM THE PROTOCOL

We will not summarize smoking and alcohol use as baseline characteristics.

## 9. DATA NOT SUMMARISED OR PRESENTED

Not applicable in the study.

#### 10. REFERENCES

1. C Garnett, K Needleman, J Liu, R Brundage and Y Wang. Operational Characteristics of Linear Concentration-QT Models for Assessing QTc Interval in the Thorough QT and Phase I Clinical Studies. Clinical Pharmacology & Therapeutics, 2016;100(2): 120-178.

## 11. VALIDATIONS

SAS® for Windows (release 9.2 or a later version) will be used for statistical analyses.

Phoenix<sup>®</sup> WinNonlin<sup>®</sup> (release 6.3 or a later version) will be used to calculate Pharmacokinetics Parameters.

The quality of statistical results will be ensured by double programming at



## 12. LISTINGS, TABLES AND FIGURES

## 12.1 Listings

| No. | Title of listing | Analysis<br>Population/Dataset |
|---|---|---|
| 16.2.1 – Su | bject Disposition | |
| | Randomization Details | All Subjects |
| | Subject Disposition | All Subjects |
| | Analysis Population | All Subjects |
| 16.2.2 – Inc | clusion and Exclusion Criteria | |
| | Inclusion and Exclusion Criteria | All Subjects |
| 16.2.3 – De | emography and Baseline Characteristics | |
| | Demography | All Subjects |
| | Baseline Characteristics | All Subjects |
| 16.2.4 – Mo | edical History and medications | |
| | Medical history | All Subjects |
| | Prior and Concomitant Medications | All Subjects |
| 16.2.5 – Ex | posure and Compliance | |
| | Study Drug Exposure and Compliance | All Subjects |
| 16.2.6 – Ph | armacokinetics | |
| | Blood Collection Time for Pharmacokinetic Evaluation | All Subjects |
| | Plasma Concentrations | All Subjects |
| | Plasma Pharmacokinetic Parameters - Non-Compartmental | All Subjects |
| | Analysis | |
| | Plasma Pharmacokinetic Parameters - Compartmental Analysis | All Subjects |
| 16.2.7 – Ad | lverse Events | |
| | Adverse Events | All Subjects |
| 16.2.8 – Ro | outine safety laboratory tests Parameters | |
| | Routine Safety Laboratory tests - Hematology | All Subjects |
| | Routine Safety Laboratory tests - Biochemistry | All Subjects |
| | Routine Safety Laboratory tests - Coagulation | All Subjects |
| | Routine Safety Laboratory tests - Urinalysis | All Subjects |
| | Routine Safety Laboratory tests – Urinary Sediment | All Subjects |
| | Routine Safety Laboratory tests – Overall Evaluation | All Subjects |
| 16.2.9 – Ot | ther Safety assessments | <u></u> |
| | Physical Examinations, Body weight and BMI | All Subjects |
| | Vital Signs | All Subjects |
| | Routine Safety 12-Lead ECG | All Subjects |

## 12.2 Tables

| No. Title of table | Analysis Population/Dataset |
|----------------------|-----------------------------|
| 14.1 – Study | |
| Subjects Disposition | All Subjects |

| No. | Title of table | Analysis<br>Population/Dataset |
|---|---|---|
| <u> 81 (Abril 19-20) 74</u> | Analysis Population | All Subjects |
| | Demographics and Baseline Characteristics | Safety, PK |
| | Summary of Prior and Concomitant Medications | Safety |
| 14.2 – Ph | armacokinetics | |
| | Descriptive Statistics for Plasma Concentrations | PK |
| | Descriptive Statistics for Plasma Pharmacokinetic Parameters -<br>Non-Compartmental Analysis | PK |
| | Descriptive Statistics for Plasma Pharmacokinetic Parameters -<br>Compartmental Analysis | PK |
| 14.3 – Sa | fety | |
| | Summary of Treatment Emergent Adverse Events | Safety |
| | Treatment Emergent Adverse Events by System Organ Class and Preferred Term | Safety |
| | Treatment Emergent Adverse Events by System Organ Class,<br>Preferred Term and Severity | Safety |
| | Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Relation to Study Drug | Safety |
| | Summary of Routine safety laboratory tests - Hematology | Safety |
| | Summary of Routine safety laboratory tests - Biochemistry | Safety |
| | Summary of Routine safety laboratory tests - Coagulation | Safety |
| | Summary of Routine safety laboratory tests - Urinalysis | Safety |
| | Summary of Routine safety laboratory tests - Overall Evaluation | Safety |
| | Shift table of Routine safety laboratory tests - Urinalysis | Safety |
| | Body weight | Safety |
| | Vital Signs | Safety |
| | Vital Signs - Overall Evaluation | Safety |
| | Routine Safety 12-Lead ECG | Safety |
| | Routine Safety 12-Lead ECG - Overall Evaluation | Safety |
| | Routine Safety 12-Lead ECG - Number of Subject Meeting QTcF Criteria | Safety |

# 12.3 Figures

| No. Title of figure | Analysis Population/Dataset |
|---|---|
| 14.2 – Pharmacokinetics | |
| Profile of Mean Plasma Concentrations – PK | PK |
| Profile of Mean observed and predicted Plasma Concentrations - Compartmental Analysis - PK | PK |
| 16.2.6 – Pharmacokinetics | |
| Profile of Individual observed and predicted Plasma Concentrations by Subjects - Compartmental Analysis | PK |

| No. | Title of figure | Analysis<br>Population/Dataset |
|---|---|---|
| | Profile of Individual observed Plasma Concentrations by Each | PK |
| | Group | |

## 13. REVISION HISTORY FOR SAP AMENDMENTS

Version 2.0 (25 January, 2019)

It reflected the results of the data review meeting on 17 January, 2019.

In List of PK Parameters, the PK parameters were matched with those described in PK Parameter Calculations in Appendix 1 and 2.

In Section 1, description of Section 3 has been deleted because Holter ECG analysis was not described.

At the beginning of Section 2, "In this SAP, the analyses with underline are not planed." was added, and the contents of analysis in Section 2.1.1, 2.1.3 and 2.1.4 were underlined.

# APPENDIX 1 – CALCULATION OF PHARMACOKINETIC PARAMETER USING NON-COMPARTMENTAL ANALYSIS

- Actual blood sampling times for the assay of MCI-186 will be used in the calculation of pharmacokinetic parameters
- All concentrations below the LLOQ will be set at zero for pharmacokinetic calculations
- Calculation of pharmacokinetic parameters will be used 1/Y weighting of the data
- When  $\lambda_z$  is missing (or cannot be determined), AUC<sub>0-\infty</sub>, AUC%<sub>ex</sub>, MRT, CL, V<sub>ss</sub>, V<sub>z</sub>, Lower limited of  $\lambda_z$ , Upper limited of  $\lambda_z$  and Number of  $\lambda_z$  points will not be calculated

| PK Parameter Calculations | | |
|---|---|---|
| Parameters | Unit | Calculation |
| AUC <sub>0-last</sub> | h•ng/mL | will be calculated using the linear trapezoidal method and actual times $AUC_{0-last} = \sum_{i=1}^n \frac{t_i - t_{i-1}}{2} \left( C_{i-1} + C_i \right)$ |
| AUC <sub>0-24h</sub> | h•ng/mL | will be calculated using the linear trapezoidal method and zero to 24h of actual times |
| AUC <sub>0-∞</sub> | h•ng/mL | $AUC_{0-\infty} = AUC_{0-last} + \frac{C_{last}}{\lambda_{z}}$ |
| AUC% <sub>ex</sub> | % | $AUC\%_{ex} = \frac{AUC_{0-\infty} - AUC_{0-last}}{AUC_{0-\infty}} \times 100$ |
| C <sub>max</sub> | ng/mL | will be determined using maximum drug concentration |
| CL | L/h | $CL = \frac{Dose}{AUC_{0-\infty}}$ |

| Parameters | Unit | Calculation |
|---|---|---|
| $\lambda_z$ | 1/h | The exponential rate constant of the terminal phase, $\lambda_z$ , will be estimated by log-linear regression, if determinable. The number of data points included in the regression will be determined by visual inspection. Wherever possible, a minimum of 3 data points will be used in the estimation of $\lambda_z$ . |
| | | During the analysis, this calculation method repeats regressions using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to $C_{max}$ or prior to the end of infusion will not be used unless the user specifically requests that time range. Points with a value of zero for the dependent variable will be excluded. For each regression, an adjusted $R^2$ will be computed |
| | | Adjusted R <sup>2</sup> = $1 - \frac{(1 - R^2) + (n - 1)}{(n - 2)}$ |
| | | where n is the number of data points in the regression and $R^2$ is the square of the correlation coefficient. |
| | | The regression with the largest adjusted R <sup>2</sup> will be selected to |
| | | estimate $\lambda_z$ , with these caveats: |
| | | If the adjusted $R^2$ does not improve, but is within 0.0001 of the largest adjusted $R^2$ value, the regression with the larger number of points will be used. $\lambda_z$ must be positive, and calculated from at least three data points. |
| Lower limited of $\lambda_z$ | h | will be determined using lower limit on time to be included in the calculation of $\lambda_z$ |
| MRT | h | $AUMC_{0-\infty} = \sum_{i=1}^{n} \frac{(t_i - t_{i-1})(t_i \times C_i + t_{i-1} \times C_{i-1})}{2} + \frac{t \times C_t}{\lambda_z} + \frac{C_t}{(\lambda_z)^2}$ |
| | | $MRT = \frac{AUMC_{0-\infty}}{AUC_{0-\infty}} - \frac{TI}{2}$ where TI represents infusion duration. |
| Number of $\lambda_z$ points | - | will be determined using number of points used in computing $\lambda_z$ . If $\lambda_z$ cannot be estimated, zero. |
| t <sub>1/2</sub> | h | $t_{1/2}$ will be determined as: $t_{1/2} = \frac{\log_e(2)}{\lambda_2}$ |

| PK Parameter Calculations | | |
|---|---|---|
| Parameters | Unit | Calculation |
| t <sub>max</sub> | h | will be determined using time to maximum drug concentration |
| Upper limited of $\lambda_z$ | h | will be determined using upper limit on time to be included in the calculation of $\lambda_{z}$ |
| V <sub>ss</sub> | L | $V_{ss} = MRT \times CL$ |
| V <sub>z</sub> | L | $V_z = CL \times \frac{1}{\lambda_z}$ |

# APPENDIX 2 – CALCULATION OF PHARMACOKINETIC PARAMETER USING COMPARTMENTAL ANALYSIS

- Actual blood sampling times for the assay of MCI-186 will be used in the calculation of pharmacokinetic parameters.
- All concentrations below the LLOQ will be set at missing for pharmacokinetic calculations.
- In this model, use the three-compartment model as shown in the figure.



- Plasma concentration formula in infusion  $(0 \le t \le T)$  is as follows.

$$Cp(t) = \frac{A(1-e^{-\alpha t})}{\alpha T} + \frac{B\left(1-e^{-\beta t}\right)}{\beta T} + \frac{C(1-e^{-\gamma t})}{\gamma T}$$

Plasma concentration formula after the end of infusion  $(T \le t)$  is as follows.

$$Cp(t) = \frac{A \left(1 - e^{-\alpha T}\right)}{\alpha T} e^{-\alpha (t-T)} + \frac{B \left(1 - e^{-\beta T}\right)}{\beta T} e^{-\beta (t-T)} + \frac{C \left(1 - e^{-\gamma T}\right)}{\gamma T} e^{-\gamma (t-T)}$$

A, B and C are coefficients which describe the exponential functions of each phase  $\alpha$ ,  $\beta$  and  $\gamma$  are exponents which describe the shape of the curve for each phase

| WinNonlin PK Parameter Calculation Settings | |
|---|---|
| Model Selection | Model 19 |
| | (Three-compartment, IV-infusion, and first-order elimination rate without lag time model) |
| Mappings | Subject id, Dose, Time, Concentration |
| Weighting | 1/Yhat |
| Parameter Options | WinNonlin Generated Initial Parameter Values / WinNonlin Bounds |
| Minimization | Gauss-Newton (Levenberg and Hartley) |
| Increment for Partial Derivatives | 0.001 |

| WinNonlin PK Parameter Calculation Settings | |
|---------------------------------------------|--------|
| Meansquare | |
| Iterations | 50 |
| Convergence criteria | 0.0001 |

| | | PK Parameter Calculations |
|---|---|---|
| Parameters | Unit | Calculation |
| A | ng/mL | $A = \frac{D(k_{21} - \alpha)(k_{31} - \alpha)}{V_1(\gamma - \alpha)(\beta - \alpha)}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |
| В | ng/mL | $B = \frac{D(k_{21} - \beta)(k_{31} - \beta)}{V_1(\gamma - \beta)(\alpha - \beta)}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |
| C | ng/mL | $C = \frac{D(k_{21} - \gamma)(k_{31} - \gamma)}{V_1(\alpha - \gamma)(\beta - \gamma)}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |
| α | 1/h | $\alpha = \frac{\mathbf{k_{21} \cdot k_{31} \cdot k_{el}}}{\beta \cdot \gamma}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |
| β | 1/h | $\beta = \frac{\mathbf{k_{21} \cdot k_{31} \cdot k_{el}}}{\alpha \cdot \gamma}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |
| γ | 1/h | $\gamma = \frac{\mathbf{k_{21} \cdot k_{31} \cdot k_{el}}}{\alpha \cdot \beta}$ |
| | | An initial value is obtained from the above relational formula, and an estimated value is calculated using a nonlinear least squares method. |

| PK Parameter Calculations | | |
|---|---|---|
| Parameters | Unit | Calculation |
| $V_1$ | L | $V_1 = \frac{D}{A + B + C}$ |
| $k_{\rm el}$ | 1/h | $k_{el} = \frac{CL}{V_1}$ |
| k <sub>21</sub> | 1/h | $k_{21} = \frac{\alpha \cdot \beta \cdot \gamma}{k_{el} \cdot k_{31}}$ |
| k <sub>31</sub> | 1/h | $k_{31} = \frac{\alpha \cdot \beta \cdot \gamma}{k_{el} \cdot k_{21}}$ |
| C <sub>max</sub> | ng/mL | will be determined using maximum drug concentration |
| t <sub>1/2α</sub> | h | $t_{1/2\alpha} = \frac{\ln(2)}{\alpha}$ |
| t <sub>1/2β</sub> | h | $t_{1/2\beta} = \frac{\ln(2)}{\beta}$ |
| t <sub>1/2γ</sub> | h | $t_{1/2\gamma} = \frac{\ln(2)}{\gamma}$ |
| AUC <sub>0-∞</sub> | h•ng/mL | $AUC_{0-\infty} = \frac{A}{\alpha} + \frac{B}{\beta} + \frac{C}{\gamma}$ |
| CL | L/h | $CL = \frac{D}{AUC_{0-\infty}}$ |
| MRT | h | $AUMC = \frac{A}{\alpha} \left( \frac{T}{2} + \frac{1}{\alpha} \right) + \frac{B}{\beta} \left( \frac{T}{2} + \frac{1}{\beta} \right) + \frac{C}{\gamma} \left( \frac{T}{2} + \frac{1}{\gamma} \right)$ |
| | | $MRT = \frac{AUMC}{AUC_{0-\infty}}$ |
| $V_{SS}$ | L | $V_{SS} = CL \cdot MRT$ |